CLINICAL TRIAL: NCT00127764
Title: European Randomised Placebo-Controlled Trial of Adjuvant Oral Glucocorticoid Pulse Therapy in Pemphigus (Pempuls Trial)
Brief Title: European Trial of Adjuvant Oral Glucocorticoid Pulse Therapy in Pemphigus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 754309
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2004-08

CONDITIONS: Pemphigus
Keywords: pemphigus; dexamethasone; glucocorticoids; pulse; therapy; randomised; placebo-controlled
MeSH Terms: conditions — Pemphigus | interventions — Dexamethasone

INTERVENTIONS:
Drug: dexamethasone (50mg 1dd6, 3 consecutive days/month)

SUMMARY:
By this study, the investigators want to test if the value of adjuvant pulse glucocorticoid therapy for pemphigus can be determined by comparing an experimental arm (dexamethasone pulse therapy, prednisolone, and azathioprine) with a control arm (placebo pulse therapy, prednisolone, and azathioprine). The investigators will determine the rate of complete remission with dexamethasone pulse therapy; the time needed for complete remission; and the duration of remission, and compare these data with those of the placebo arm.

DETAILED DESCRIPTION:
Pemphigus is a severe chronic dermatological disease which appears to be incurable. Oral glucocorticoid now forms the cornerstone of treatment. From previous uncontrolled studies it has been suggested, that the use of high dose intravenous glucocorticoid pulse therapy may lead to complete remission without further therapy. Prospective placebo-controlled studies of adjuvant pulse therapy for pemphigus are lacking. This prospective, multi-centre, randomised, double-blind, placebo-controlled trial assesses the efficacy and steroid-sparing effect of oral high-dose glucocorticoid pulse therapy as adjuvant added to the standard combination therapy of prednisone and azathioprine in the treatment of pemphigus vulgaris, in terms of complete remission rate (primary endpoint), initial control, disease control, and adverse events. In the experimental arm glucocorticoid pulse therapy is given, comprising monthly pulses with 300mg oral dexamethasone on three consecutive days. In addition the patients receive daily prednisone and azathioprine treatment, the latter dose adjusted to the thiopurine-methyltransferase level. In the control arm the glucocorticoid pulse therapy is replaced double blindly by monthly oral placebo capsules on three consecutive days. in addition the patients receive the same daily combination schedule with prednisone and azathioprine as in the experimental arm. This study design requires 30 patients in each arm, with one year follow-up. Only new patients with pemphigus vulgaris and/or pemphigus oris are included.

ELIGIBILITY:
Inclusion Criteria:

* New patients with diagnosis of pemphigus vulgaris

Exclusion Criteria:

* Diagnosis of pemphigus different from vulgaris type
* Current use of adjuvant treatment other than azathioprine. A wash out period of at least 2 weeks is required before inclusion is acceptable.
* Presence of contra-indications for the use of high dose steroids
* No availability for follow-up.
* Concomitant diseases treated with oral steroids.
* Glucocorticoids administered for pemphigus vulgaris longer than two months.
* Presence of contra-indications for the use of azathioprine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-01; Study Completion 2005-04

PRIMARY OUTCOMES:
The rate of complete remission with pulse therapy
Number of weeks in complete remission after 12 months

SECONDARY OUTCOMES:
Time from start of pulse therapy until initial control
Number of weeks in remission until 12 months
Cumulative prednisolone use until 12 months
Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Marcel F Jonkman, MD, PhD, Principal Investigator — Department of Dermatology, University Medical Center Groningen
Locations (1):
- Department of Dermatology, University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Toth GG, van de Meer JB, Jonkman MF. Dexamethasone pulse therapy in pemphigus. J Eur Acad Dermatol Venereol. 2002 Nov;16(6):607-11. doi: 10.1046/j.1468-3083.2002.00413.x. PMID 12482045
- [Background] Toth GG, Westerlaken BO, Eilders M, Laseur M, Jonkman MF, Uges DR. Dexamethasone pharmacokinetics after high-dose oral therapy for pemphigus. Ann Pharmacother. 2002 Jun;36(6):1108-9. doi: 10.1345/aph.1A047. No abstract available. PMID 12058710
- [Background] Toth GG, Kloosterman C, Uges DR, Jonkman MF. Pharmacokinetics of high-dose oral and intravenous dexamethasone. Ther Drug Monit. 1999 Oct;21(5):532-5. doi: 10.1097/00007691-199910000-00007. PMID 10519450
- [Background] Toth GG, Jonkman MF. Therapy of pemphigus. Clin Dermatol. 2001 Nov-Dec;19(6):761-7. doi: 10.1016/s0738-081x(00)00190-5. No abstract available. PMID 11705686
- [Result] Mentink LF, Mackenzie MW, Toth GG, Laseur M, Lambert FP, Veeger NJ, Cianchini G, Pavlovic MD, Jonkman MF. Randomized controlled trial of adjuvant oral dexamethasone pulse therapy in pemphigus vulgaris: PEMPULS trial. Arch Dermatol. 2006 May;142(5):570-6. doi: 10.1001/archderm.142.5.570. PMID 16702494